CLINICAL TRIAL: NCT04081688
Title: A Phase I Trial of Atezolizumab and Varlilumab in Combination With Radiation in Patients With Metastatic Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Atezolizumab and Varlilumab in Combination With Radiation Therapy for NSCLC
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: accrual goal met
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Salma Jabbour, MD, Assistant Professor, Rutgers Cancer Institute of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 031912; NCI-2019-05810 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Pro2019000923; Pro2019000923 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH)
Record Dates: First submitted 2019-08-29; First posted 2019-09-09 (Actual); Results first posted 2023-06-02 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Refractory Lung Non-Small Cell Carcinoma; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — atezolizumab; Injections; Radiosurgery; varlilumab; Immunoglobulin G; Disulfides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (varlilumab, atezolizumab, SBRT) (Experimental): Patients receive varlilumab IV over 90 minutes and atezolizumab IV over 30-60 minutes every cycle. Cycles repeat every 21 days for up to 1 year (18 cycles) in the absence of disease progression or unacceptable toxicity. Between cycle 1 and 2, patients also receive SBRT.
  Interventions: Drug: Atezolizumab 1200 MG in 20 ML Injection; Radiation: Stereotactic Body Radiation Therapy; Drug: Varlilumab 3 mg/kg

INTERVENTIONS:
Drug: Atezolizumab 1200 MG in 20 ML Injection — Given IV every 3 weeks (cycle is 21 days)
  Other Names: ATEZOLIZUMAB; MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG7446; RO5541267; Tecentriq
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT between cycle 1 and cycle 2 (each cycle is 21 days)
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy
Drug: Varlilumab 3 mg/kg — Given IV every 3 weeks (cycle is 21 days)
  Other Names: CDX 1127; CDX-1127; Immunoglobulin G1, Anti-(Human CD Antigen CD27) (Human Monoclonal CDX-1127 Clone 1f5 Heavy Chain), Disulfide with Human Monoclonal CDX-1127 Clone 1f5 Kappa-chain, Dimer; VARLILUMAB

SUMMARY:
This phase I trial studies the side effects of atezolizumab, varlilumab, and radiation therapy in treating patients with non-small cell lung cancer that has spread to other places in the body (advanced) and cannot be removed by surgery (unresectable). Immunotherapy with monoclonal antibodies such as atezolizumab may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Immunotherapy with monoclonal antibodies such as varlilumab may induce changes in body?s immune system and may interfere with the ability of tumor cells to grow and spread. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Giving atezolizumab, varlilumab, and radiation therapy may increase the amount of time the disease is not active or does not spread to another part of the body.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the safety and tolerability of combined therapy with atezolizumab and varlilumab in combination with radiation in adult patients with metastatic non-small cell lung cancer (NSCLC) who have progressed on prior PD-1/PD-L1 therapy.

SECONDARY OBJECTIVES:

I. To determine objective response rate (excluding the irradiated lesion) of therapy with atezolizumab and varlilumab in combination with radiation.

II. To estimate clinical benefit rate of the combination. III. To estimate median progression-free survival of the combination. IV. To compare the frequency of immune-related adverse events (irAEs).

OUTLINE:

Patients receive varlilumab intravenously (IV) oand atezolizumab IV every 3 weeks or each cycle. Between cycle 1 and 2, patients also receive stereotactic body radiation therapy (SBRT).

After completion of study treatment, patients are followed up at 30 days, then every 3 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Must have signed and dated written informed consent form in accordance with regulatory and institutional guidelines
* Histological or cytological evidence of advanced, unresectable NSCLC
* Patients must be PD-1/PD-L1 experienced with disease progression documented either on therapy with anti-PD-1/PD-L1 or within 12 weeks of the last dose. Treatment should be initiated at least 4 weeks since last dose of PD-1/PD-L1 targeted therapy
* Patients must have progressed on at least one line of prior platinum-based chemotherapy in the metastatic setting. Subjects with unresectable stage III NSCLC who received platinum-based chemotherapy as part of chemoradiation or consolidation chemotherapy after chemoradiation are eligible if they progress within 6 months of last dose of chemotherapy. Treatment should be initiated at least 4 weeks since last dose of systemic therapy
* Subjects with an actionable molecular alteration (such as EGFR mutation, ALK or ROS1 rearrangement, BRAF V600E mutation) are eligible only after failing standard-of-care targeted therapy with tyrosine kinase inhibitor (TKI). Patients with a EGFR T790M resistant mutation must have failed a 3rd generation TKI such as osimertinib
* Must not have received any prior therapy with immune regulatory molecule (such as targeting OX-40, IDO-1, LAG-3) or anti-CD27 monoclonal antibody (including varlilumab)
* Must have at least one lesion that has not previously been irradiated (and is not within a previously radiated field) and for which palliative radiation is potentially indicated. The lesion to be irradiated must be in the lung. Patient must have at least one additional measurable lesion (other than the lesion being radiated) as per immune-related Response Evaluation Criteria in Solid Tumors (irRECIST) criteria. Patient must agree to undergo a mandatory biopsy of the non-irradiated lesion pre-treatment and post-treatment (after cycle 2). Pre-treatment tissue obtained by biopsy or resection performed according to standard of care may be utilized, provided tissue was obtained within 8 weeks of study entry, and subsequent to the last systemic anticancer therapy received
* Patients should have fewer than 10 metastatic sites and expected survival of more than 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Treatment to be initiated at least 2 weeks since last dose of prior systemic anticancer therapy (chemotherapy, radiation, and/or surgery)
* Recovery to grade 1 of any clinically significant toxicity (excluding alopecia, grade 2 fatigue, vitiligo, endocrinopathies on stable replacement therapy, grade 2 neuropathy from chemotherapy and grade 2 hearing loss from platinum chemotherapy) prior to initiation of study drugs
* Female patients of childbearing potential have a negative pregnancy test at baseline. Females of childbearing potential are defined as sexually mature women without prior hysterectomy or who have had any evidence of menses in the past 12 months. However, women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, anti-estrogens, or ovarian suppression

  * Women of childbearing potential (i.e., menstruating women) must have a negative urine pregnancy test (positive urine tests are to be confirmed by serum test) documented within 14 days of treatment initiation
  * Sexually active women of childbearing potential enrolled in the study must agree to use 2 forms of accepted methods of contraception during the course of the study and for 12 weeks after their last dose of study drug. Effective birth control includes (a) intrauterine device plus 1 barrier method; (b) on stable doses of hormonal contraception for at least 3 months (e.g., oral, injectable, implant, transdermal) plus one barrier method; (c) 2 barrier methods. Effective barrier methods are male or female condoms, diaphragms, and spermicides (creams or gels that contain a chemical to kill sperm); or (d) a vasectomized partner
  * For male patients who are sexually active and who are partners of premenopausal women: agreement to use 2 forms of contraception as in criterion above during the treatment period and for 12 weeks after the last dose of study drug
* Absolute neutrophil count >= 1,500/uL
* Platelet count >= 100,000/uL
* Hemoglobin >= 9.0 g/dL
* Total bilirubin =< 2 x upper limit of normal (ULN) or =< 3 x ULN for subjects with Gilbert?s disease or liver metastases
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN (=< 5 x ULN if evidence of hepatic involvement by malignant disease)
* Creatinine =< 1.5 x ULN or estimated glomerular filtration rate (eGFR) >= 40 mL/min/1.73m^2
* Measurable disease according to irRECIST obtained by imaging within 28 days prior to treatment initiation

Exclusion Criteria:

* Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 23 weeks (female) or 31 weeks (male) after the last dose of study drug
* Treatment with any investigational agent within 28 days prior to registration for protocol therapy
* History of psychiatric illness or social situations that would limit compliance with study requirements. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject?s participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Known active, untreated central nervous system (CNS) metastases and/or carcinomatous meningitis except for patients with =< 3 small (< 0.6 cm) asymptomatic brain lesions where treatment is not indicated. Patients with neurological symptoms must undergo a head computed tomography (CT) scan or brain magnetic resonance imaging (MRI) to exclude brain metastasis. Patients whose brain metastases have been treated may participate provided they show radiographic stability (defined as 2 brain images obtained after treatment to the brain metastases at least 4 weeks apart and show no evidence of intracranial progression)
* Known history of human immunodeficiency virus (HIV) or active hepatitis B (by surface antigen expression or polymerase chain reaction [PCR]) or active hepatitis C (by PCR) infection
* Diagnosis of immunodeficiency or is receiving systemic steroid therapy (> 10 mg daily prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to study registration
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs) or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Vitiligo, alopecia, hypothyroidism only requiring hormone replacement, psoriasis not requiring systemic treatment, celiac disease controlled by diet alone or conditions not expected to recur in the absence of an external trigger are permitted
* Documented history of a cerebral vascular event (stroke or transient ischemic attack), unstable angina, myocardial infarction, or cardiac symptoms consistent with New York Heart Association (NYHA) class III?IV within 6 months prior to their first dose of study drugs
* Prior malignancies (except non-melanoma skin cancers, and the following in situ cancers: bladder, gastric, colon, endometrial, cervical/dysplasia, melanoma, or breast) unless a complete remission was achieved at least 1 year prior to study entry
* Any active grade 3 or higher viral, bacterial, or fungal infection within 2 weeks of the first dose of the study drugs. Routine antimicrobial prophylaxis is permitted
* Active diverticulitis
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug-induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest CT scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jyoti Malhotra, Principal Investigator — Rutgers Cancer Institute of New Jersey; Salma Jabbour, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Varlilumab, Atezolizumab, SBRT)
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Varlilumab, Atezolizumab, SBRT)
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 3 and 4 Toxicity
Description: Will include grade 3 and 4 toxicities as defined by the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.
Time Frame: Up to 30 days after the last dose of treatment, an average of a year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Varlilumab, Atezolizumab, SBRT)
Number analyzed (Participants) | 15
Participants | 2

2. Secondary Outcome: To Determine Objective Response Rate (ORR) of Therapy
Description: Will be defined as the proportion of all subjected confirmed with an immune-related partial response (irPR) or immune-related complete response (irCR) divided by the number of assigned patients according to immune-related Response Evaluation Criteria in Solid Tumors (irRECIST).
Time Frame: From the start of treatment until disease progression/recurrence, assessed up to 1 year
Reporting Status: Not Posted

3. Secondary Outcome: To Estimate Clinical Benefit Rate of the Combination
Description: Will be defined as the percentage of patients who achieve irCR, irPR, and immune-related stable disease.
Time Frame: Up to 1 year
Reporting Status: Not Posted

4. Secondary Outcome: To Estimate Median Progression-free Survival (PFS) of the Combination
Description: The log-rank test will be used to analyze PFS for comparison of treatment effects, i.e., the only covariate that will be used is the treatment arm. Distributions of PFS times will be estimated using the Kaplan- Meier product-limit method. The median PFS times with two-sided 95% confidence intervals will be estimated for each treatment group.
Time Frame: From cycle 1, day 1 (each cycle is 21 days) of treatment until the criteria for disease progression is met as defined by irRECIST or death as a result of any cause, assessed up to 1 year
Reporting Status: Not Posted

5. Secondary Outcome: To Compare the Frequency of Immune-related Adverse Events (irAEs)
Description: irAE's are defined as any treatment-related AE that is inflammatory in nature, consistent with the mechanism of action of immunotherapy and generally medically manageable with topical and/or systemic immunosuppressants.
Time Frame: Up to 30 days after the last dose of treatment
Reporting Status: Not Posted

6. Other Pre Specified Outcome: To Compare Pre- and Post-treatment Tumor PD-L1 Expression
Description: Will be assessed by immunohistochemistry (IHC) and will score the percentage of cells staining positively for PD-L1 incrementally. Scoring will be performed for the percentage of malignant tumor cells and for the percentage of nonmalignant inflammatory cell compartment that express PD-L1, separately.
Time Frame: Baseline up to cycle 2, day 8 (each cycle is 21 days)
Reporting Status: Not Posted

7. Other Pre Specified Outcome: To Compare Pre- and Post-treatment Tumor Levels of Infiltrating CD3+, CD8+ T-cells
Description: Will be assessed by IHC staining to identify tumor infiltrating lymphocytes at the tumor stroma interface.
Time Frame: Baseline up to cycle 2, day 8 (each cycle is 21 days)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 30 days after the last dose of treatment, an average of a year.
Arm/Group | Treatment (Varlilumab, Atezolizumab, SBRT)
All-Cause Mortality (participants affected / at risk) | 12/15
Serious Adverse Events (participants affected / at risk) | 8/15
Other Adverse Events (participants affected / at risk) | 12/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Varlilumab, Atezolizumab, SBRT) (N=15)
Colitis (Gastrointestinal disorders) | 1 (1)
Dehydration (General disorders) | 1 (1)
Lung infestations (Injury, poisoning and procedural complications) | 3 (3)
Confusion (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Varlilumab, Atezolizumab, SBRT) (N=15)
Nausea (Gastrointestinal disorders) | 5 (7)
Lymphocyte count decreased (Investigations) | 5 (5)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pain (General disorders) | 2 (2)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 6 (10)
Hypotension (Vascular disorders) | 1 (1)
Infections and infestations (Infections and infestations) | 4 (4)
Nervous system disorders (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 1 (2)
Lipase increased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Vascular disorders (Vascular disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-06): https://cdn.clinicaltrials.gov/large-docs/88/NCT04081688/Prot_SAP_002.pdf
  • Informed Consent Form (2022-04-06): https://cdn.clinicaltrials.gov/large-docs/88/NCT04081688/ICF_000.pdf